CLINICAL TRIAL: NCT04468750
Title: The Effect of Kinesiotaping on Glenohumeral Shoulder Subluxation in Post-stroke Patients
Brief Title: Kinesiotaping Effect Glenohumeral Shoulder Subluxation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Collaborators: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5416
Record Dates: First submitted 2020-07-09; First posted 2020-07-13 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Stroke; Subluxation, Glenohumeral
MeSH Terms: conditions — Stroke; Shoulder Dislocation | interventions — Athletic Tape

STUDY DESIGN:
Intervention Model Description: This study is a quasi-experimental, single-subject AB design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Kinesiotape (Experimental): Kinesiotape (Nasara, Korea) was applied for three times a week (Monday, Wednesday, and Friday) for three weeks.
  Interventions: Device: kinesiotape

INTERVENTIONS:
Device: kinesiotape — During the rehabilitation program, all patients with GHS had kinesiotaping three times a week.

SUMMARY:
To evaluate the effectiveness of the kinesiotaping on pain, recovery of movement and daily life activities in Turkish hemiplegic patients.

ELIGIBILITY:
Inclusion Criteria:

* (1) 18 to 90 years of age, (2) stroke onset within one year, (3) shoulder subluxation in the involved upper extremity and (4) being oriented and cooperative.

Exclusion Criteria:

* (1) global aphasia, (2) malignancy, (3) previous shoulder pain or surgery, (4) other neuromuscular disorders and (5) severe cardiopulmonary disease that affects daily life activities.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-11-13 (Actual); Primary Completion 2015-07-15 (Actual); Study Completion 2018-06-06 (Actual)

PRIMARY OUTCOMES:
Subluxation degree by physical examination | 0-3weeks
  A clinician measured the gap between the acromion and the humeral head with the fingerbreadth at the distal interphalangeal joint of the right index and middle fingers
Subluxation degree by radiograph | 0-3weeks
  The anterio-posterior shoulder X-ray was taken in an erect position, and subluxation was evaluated by Van Langenberghe's five point classification.
physical examination | 0-3weeks
  Passive range of motion (Flexion and Abduction)

SECONDARY OUTCOMES:
Evaluation of the pain of the shoulder | 0-3weeks
  Pain with motion was measured by a verbal descriptive pain scale. The VDPS was developed by Melzack and Katz and is composed of words such as "mild" (level 1) to "very severe pain" (level 5)
Evaluation of Daily life activities | 0-3weeks
  Daily life activities were evaluated using the Katz index of independence in activities of daily living, which evaluates the patients in bathing, dressing, toileting, transferring, continence, and eating. Activities were scored as zero or one with the total score ranging from zero to six. Higher scores are related with higher independency.

CONTACTS AND LOCATIONS:
Overall Officials: Halil Ucan, MD, Study Director — Ankara Physical Medicine and Rehabilitation Education and Research Hospital

IPD SHARING:
Plan to Share IPD: No